CLINICAL TRIAL: NCT02806908
Title: A Randomized, Double-Blind, Placebo-Controlled, Crossover On-Road Driving Study Assessing the Effect of JZP-110 on Driving Performance in Subjects With Excessive Sleepiness Due to Narcolepsy
Brief Title: Study Assessing Effects of JZP-110 on Driving Performance in the Treatment of Excessive Sleepiness in Narcolepsy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 15-005
Record Dates: First submitted 2016-06-10; First posted 2016-06-21 (Estimated); Results first posted 2021-01-13 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2020-12

CONDITIONS: Narcolepsy; Excessive Sleepiness
Keywords: Driving
MeSH Terms: conditions — Narcolepsy; Disorders of Excessive Somnolence | interventions — solriamfetol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Once daily dosing
  Interventions: Drug: Placebo
- JZP-110 (Active Comparator): 150 mg/day for first 3 days and 300 mg/day for next 4 days
  Interventions: Drug: JZP-110

INTERVENTIONS:
Drug: JZP-110
  Other Names: solriamfetol
  Arms: JZP-110
Drug: Placebo
  Arms: Placebo

SUMMARY:
This trial is a randomized, double-blind, placebo-controlled, crossover study to evaluate the effect of JZP-110 on driving performance in subjects with excessive sleepiness due to narcolepsy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age 21 to 65 years inclusive
2. Diagnosis of narcolepsy per International Classification of Sleep Disorders (ICSD-3) or Diagnostic and Statistical Manual of Mental Disorders 5th Edition (DSM-5)
3. BMI 18 to <40 kg/m2
4. Willing and able to provide written informed consent

Exclusion Criteria:

1. Female subjects who are pregnant, nursing, or lactating
2. Moderate or severe sleep apnea
3. Any other clinically relevant medical, behavioral, or psychiatric disorder other than narcolepsy that is associated with excessive sleepiness
4. History or presence of bipolar disorder, bipolar related disorders, schizophrenia, schizophrenia spectrum disorders, or other psychotic disorders according to DSM-5 criteria
5. History or presence of any unstable medical condition, behavioral or psychiatric disorder (including active suicidal ideation), or surgical history that could affect the safety of the subject or interfere with study efficacy and/or safety assessments per the judgment of the investigator
6. History of bariatric surgery within the past year or a history of any gastric bypass procedure
7. Presence or history of significant cardiovascular disease
8. Unable to washout or refrain from taking any over-the-counter (OTC) or prescription medications that could affect sleep-wake function

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-06; Primary Completion 2019-05-19 (Actual); Study Completion 2019-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grace Wang, MD, Study Director — Jazz Pharmaceuticals; Jan Ramaekers, PhD, Principal Investigator — Maastricht University
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] Devine JK, Schwartz L, Hursh S, Asin J, de Vries N, Vonk PE, Vermeeren A, Donjacour CEHM, Vinckenbosch F, Ramaekers JG, Janssen H, Wang G, Chen D, Carter LP, Overeem S, Lammers GJ. Psychomotor Vigilance Performance in Participants with Excessive Daytime Sleepiness in Obstructive Sleep Apnea or Narcolepsy Compared with SAFTE-FAST Model Predictions. Neurol Ther. 2023 Feb;12(1):249-265. doi: 10.1007/s40120-022-00425-w. Epub 2022 Dec 10. PMID 36494591

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo/JZP-110: Subjects received Placebo for 7 days or JZP-110 (150 mg/day for 3 days, followed by 300 mg/day for 4 days) in a counterbalanced order between Treatment Period 1 and Treatment Period 2.
- JZP-110/Placebo: Subjects received JZP-110 (150 mg/day for 3 days, followed by 300 mg/day for 4 days) or the matching placebo for 7 days in a counterbalanced order between Treatment Period 1 and Treatment Period 2.
Period: Overall Study
Arm/Group | Placebo/JZP-110 | JZP-110/Placebo
Started | 11 | 13
Completed | 10 | 12
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- JZP-110/Placebo: JZP-110 (150 mg/day for 3 days, followed by 300 mg/day for 4 days) or the matching placebo for 7 days in Treatment Period 1 or Treatment Period 2.
- Total: Total of all reporting groups
Arm/Group | Placebo/JZP-110 | JZP-110/Placebo | Total
Number analyzed (Participants) | 11 | 13 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.2 (10.81) | 41.4 (13.00) | 40.4 (11.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 6 | 7 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 9 | 12 | 21
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Netherlands | 11 | 13 | 24

OUTCOME MEASURES:

1. Primary Outcome: Standard Deviation of Lateral Position (SDLP) at 2 Hours Post-dose (Approximately at Tmax)
Description: Subjects were instructed to drive with steady lateral position between the delineated boundaries of the slower (right) traffic lane, while maintaining a constant speed of 95 kilometers (km) per hour (hr). Deviation was measured by the vehicle's speed and lateral distance to the left lane line and was continuously recorded. Individual improvement was defined as a decrease in SDLP below the negative value of threshold; individual impairment was defined as an increase in SDLP above the threshold or failure to complete the driving test due to sleepiness or subjects related safety concerns.
Time Frame: 2 hours post-dose
Population: The modified intent to treat (mITT) population consisted of 22 subjects.
Measure: Median (Full Range); unit: centimeter (cm)
Groups:
- Placebo: Subjects received a single oral daily dose of placebo for 7 days in Treatment Period 1 or Treatment Period 2 in a counterbalanced order.
- JZP-110: Subjects received a single oral daily dose of JZP-110 (150 mg/day for 3 days) then JZP-110 (300 mg/day for 4 days) during Treatment Period 1 or Treatment Period 2 in a counterbalanced order.
Arm/Group | Placebo | JZP-110
Number analyzed (Participants) | 22 | 22
centimeter (cm) | 20.46 [14.4 to 28.6] | 19.08 [13.2 to 25.0]
Statistical Analysis 1: Comparison: Placebo vs JZP-110; Test type: Superiority; p = 0.0022, ANOVA

2. Secondary Outcome: SDLP at 6 Hours Post-dose
Description: as for outcome 1
Time Frame: 6 hours post-dose
Population: Subjects in the modified intent-to-treat (mITT) population who did not have an assessment for a particular endpoint were excluded in the analysis of that endpoint.
Measure: Median (Full Range); unit: cm
Arm/Group | Placebo | JZP-110
Number analyzed (Participants) | 21 | 22
cm | 19.78 [14.6 to 38.9] | 19.59 [13.0 to 26.9]
Statistical Analysis 1: Comparison: Placebo vs JZP-110; Test type: Superiority; p = 0.0416, ANOVA

3. Secondary Outcome: Number of Subjects With Improved or Impaired Driving at a Threshold 1 Centimeter (cm) on JZP-110 Compared to Placebo 2 Hours Post-dose
Description: Individual changes (solriamfetol minus placebo) in driving performance were measured by SDLP at 2 hours postdose. The Maximum McNemar symmetry analyses was used to detect an asymmetry in the distribution of the change in driving performance at 2 hours postdose. The test examined the differences in the proportions of impaired drivers and improved drivers following treatment using a generalized single McNemar test statistics were obtained at each threshold (1.0, 1.5, 2.0, 2.5, 3.0, and 3.5 cm), which was the vehicle weaving amount. Changes in SDLP exceeding 2.4 cm have been evaluated as clinically relevant. Improvement was defined as a decrease in SDLP comparing JZP-110 and placebo below the threshold and impairment was defined as an increase in SDLP above the threshold or failure to complete the driving test due to sleepiness or subjects related safety concerns.
Time Frame: 2 hours post-dose
Population: The arms/group titles are combined as (solriamfetol minus placebo) for this outcome measure. Pre-specified McNemar test results were defined by driving study completion status per participant as impaired or improved (JZP-110 minus Placebo). The modified intent-to-treat (mITT) analysis population was comprised of all randomized subjects who received at least one dose of study medication and had evaluable SDLP data at 2 hours postdose in any post-baseline visit.
Measure: Count of Participants; unit: Participants
Groups:
- Difference (JZP-110 -Placebo): JZP-110 - Subjects received a single oral daily dose of JZP-110 (150 mg/day for 3 days) then JZP-110 (300 mg/day for 4 days) during Treatment Period 1 or Treatment Period 2 in a counterbalanced order.
  Placebo - Subjects received a single oral daily dose of placebo for 7 days in Treatment Period 1 or Treatment Period 2 in a counterbalanced order.
Arm/Group | Difference (JZP-110 -Placebo)
Number analyzed (Participants) | 22
Participants
  Improved | 5
  Impaired | 5
Statistical Analysis 1: Comparison: Difference (JZP-110 -Placebo); Test type: Superiority; p = 0.0963, McNemar

4. Secondary Outcome: Number of Subjects With Improved or Impaired Driving at a Threshold 1.5 cm on JZP-110 Compared to Placebo 2 Hours Post-dose
Description: as for outcome 3
Time Frame: 2 hours post-dose
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Difference (JZP-110 -Placebo)
Number analyzed (Participants) | 22
Participants
  Improved | 10
  Impaired | 5
Statistical Analysis 1: Comparison: Difference (JZP-110 -Placebo); Test type: Superiority; p = 0.3018, McNemar

5. Secondary Outcome: Number of Subjects With Improved or Impaired Driving at a Threshold 2.0 cm on JZP-110 Compared to Placebo 2 Hours Post-dose
Description: as for outcome 3
Time Frame: 2 hours post-dose
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Difference (JZP-110 -Placebo)
Number analyzed (Participants) | 22
Participants
  Improved | 9
  Impaired | 5
Statistical Analysis 1: Comparison: Difference (JZP-110 -Placebo); Test type: Superiority; p = 0.4240, McNemar

6. Secondary Outcome: Number of Subjects With Improved or Impaired Driving at a Threshold 2.5 cm on JZP-110 Compared to Placebo 2 Hours Post-dose
Description: as for outcome 3
Time Frame: 2 hours post-dose
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Difference (JZP-110 -Placebo)
Number analyzed (Participants) | 22
Participants
  Improved | 6
  Impaired | 4
Statistical Analysis 1: Comparison: Difference (JZP-110 -Placebo); Test type: Superiority; p = 0.7539, McNemar

7. Secondary Outcome: Number of Subjects With Improved or Impaired Driving at a Threshold 3.0 cm on JZP-110 Compared to Placebo 2 Hours Post-dose
Description: as for outcome 3
Time Frame: 2 hours post-dose
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Difference (JZP-110 -Placebo)
Number analyzed (Participants) | 22
Participants
  Improved | 6
  Impaired | 4
Statistical Analysis 1: Comparison: Difference (JZP-110 -Placebo); Test type: Superiority; p = 0.7539, McNemar

8. Secondary Outcome: Number of Subjects With Improved or Impaired Driving at a Threshold 3.5 cm on JZP-110 Compared to Placebo 2 Hours Post-dose
Description: as for outcome 3
Time Frame: 2 hours post-dose
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Difference (JZP-110 -Placebo)
Number analyzed (Participants) | 22
Participants
  Improved | 4
  Impaired | 4
Statistical Analysis 1: Comparison: Difference (JZP-110 -Placebo); Test type: Superiority; p = 1.0000, McNemar

9. Secondary Outcome: Number of Subjects With Improved or Impaired Driving at a Threshold 1 cm on JZP-110 Compared to Placebo 6 Hours Post-dose
Description: Individual changes (solriamfetol minus placebo) in driving performance were measured by SDLP at 6 hours postdose. The Maximum McNemar symmetry analyses was used to detect an asymmetry in the distribution of the change in driving performance at 6 hours postdose. The test examined the differences in the proportions of impaired drivers and improved drivers following treatment using a generalized single McNemar test statistics were obtained at each threshold (1.0, 1.5, 2.0, 2.5, 3.0, and 3.5 cm), which was the vehicle weaving amount. Changes in SDLP exceeding 2.4 cm have been evaluated as clinically relevant. Improvement was defined as a decrease in SDLP comparing JZP-110 and placebo below the threshold and impairment was defined as an increase in SDLP above the threshold or failure to complete the driving test due to sleepiness or subjects related safety concerns.
Time Frame: 6 hours post-dose
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Difference (JZP-110 -Placebo)
Number analyzed (Participants) | 22
Participants
  Improved | 10
  Impaired | 7
Statistical Analysis 1: Comparison: Difference (JZP-110 -Placebo); Test type: Superiority; p = 0.6291, McNemar

10. Secondary Outcome: Number of Subjects With Improved or Impaired Driving at a Threshold 1.5 cm on JZP-110 Compared to Placebo 6 Hours Post-dose
Description: as for outcome 9
Time Frame: 6 hours post-dose
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Difference (JZP-110 -Placebo)
Number analyzed (Participants) | 22
Participants
  Improved | 8
  Impaired | 7
Statistical Analysis 1: Comparison: Difference (JZP-110 -Placebo); Test type: Superiority; p = 1.0000, McNemar

11. Secondary Outcome: Number of Subjects With Improved or Impaired Driving at a Threshold 2.0 cm on JZP-110 Compared to Placebo 6 Hours Post-dose
Description: as for outcome 9
Time Frame: 6 hours post-dose
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Difference (JZP-110 -Placebo)
Number analyzed (Participants) | 22
Participants
  Improved | 8
  Impaired | 7
Statistical Analysis 1: Comparison: Difference (JZP-110 -Placebo); Test type: Superiority; p = 1.0000, McNemar

12. Secondary Outcome: Number of Subjects With Improved or Impaired Driving at a Threshold 2.5 cm on JZP-110 Compared to Placebo 6 Hours Post-dose
Description: as for outcome 9
Time Frame: 6 hours post-dose
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Difference (JZP-110 -Placebo)
Number analyzed (Participants) | 22
Participants
  Improved | 8
  Impaired | 7
Statistical Analysis 1: Comparison: Difference (JZP-110 -Placebo); Test type: Superiority; p = 1.0000, McNemar

13. Secondary Outcome: Number of Subjects With Improved or Impaired Driving at a Threshold 3.0 cm on JZP-110 Compared to Placebo 6 Hours Post-dose
Description: as for outcome 9
Time Frame: 6 hours post-dose
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Difference (JZP-110 -Placebo)
Number analyzed (Participants) | 22
Participants
  Improved | 7
  Impaired | 5
Statistical Analysis 1: Comparison: Difference (JZP-110 -Placebo); Test type: Superiority; p = 0.7744, McNemar

14. Secondary Outcome: Number of Subjects With Improved or Impaired Driving at a Threshold 3.5 cm on JZP-110 Compared to Placebo 6 Hours Post-dose
Description: as for outcome 9
Time Frame: 6 hours post-dose
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Difference (JZP-110 -Placebo)
Number analyzed (Participants) | 22
Participants
  Improved | 6
  Impaired | 6
Statistical Analysis 1: Comparison: Difference (JZP-110 -Placebo); Test type: Superiority; p = 0.7539, McNemar

15. Secondary Outcome: Standard Deviation of Speed (SDS) at 2 Hours Post-dose
Description: Mean SDS was a common measure of the driver's ability to maintain a constant driving speed. Variations in driving speed were recorded and analyzed.
Time Frame: 2 hours post-dose
Measure: Least Squares Mean (Standard Error); unit: kilometers/hour (km/hr)
Arm/Group | Placebo | JZP-110
Number analyzed (Participants) | 22 | 22
kilometers/hour (km/hr) | 2.97 (0.151) | 2.76 (0.151)
Statistical Analysis 1: Comparison: Placebo vs JZP-110; Test type: Superiority; p = 0.1141, ANOVA

16. Secondary Outcome: SDS at 6 Hours Post-dose
Description: as for outcome 15
Time Frame: 6 hours post-dose
Population: Subjects in the mITT population who did not have an assessment for a particular endpoint were excluded in the analysis of that endpoint.
Measure: Least Squares Mean (Standard Error); unit: km/hr
Arm/Group | Placebo | JZP-110
Number analyzed (Participants) | 21 | 22
km/hr | 3.18 (0.153) | 3.08 (0.151)
Statistical Analysis 1: Comparison: Placebo vs JZP-110; Test type: Superiority; p = 0.4441, ANOVA

17. Secondary Outcome: Number of Lapses in Driving Test at 2 Hours Post-dose
Description: Number of driving lapses (also known as lane drift, was defined as deviations > 100 cm from the mean lateral position and from the absolute lateral position for 8 seconds. Driving performance will be assessed using a standardized on-road driving test on Day 7 (Visit 4) and on Day 14 (Visit 5). A practice driving test will be done during the screening period to familiarize the subject with the vehicle and test scenario, assess if the subject can adequately operate the manual transmission vehicle, and determine if any safety concerns exist that exclude the subject from participating in the study.
Time Frame: 2 hours post-dose
Measure: Least Squares Mean (Standard Error); unit: number of lapses
Arm/Group | Placebo | JZP-110
Number analyzed (Participants) | 22 | 22
number of lapses | 3.26 (0.834) | 2.27 (0.834)
Statistical Analysis 1: Comparison: Placebo vs JZP-110; Test type: Superiority; p = 0.3423, ANOVA

18. Secondary Outcome: Number of Lapses in Driving Test at 6 Hours Post-dose
Description: as for outcome 17
Time Frame: 6 hours post-dose
Population: as for outcome 16
Measure: Least Squares Mean (Standard Error); unit: number of lapses
Arm/Group | Placebo | JZP-110
Number analyzed (Participants) | 21 | 22
number of lapses | 3.72 (0.844) | 3.64 (0.834)
Statistical Analysis 1: Comparison: Placebo vs JZP-110; Test type: Superiority; p = 0.9384, ANOVA

19. Secondary Outcome: Psychomotor Vigilance Test (PVT) Number of Lapses at 2 Hours Post-dose
Description: The PVT was administered at screening for practice only, and at predose and within 30 minutes before each driving test on Days 7 and 14 (Visits 4 and 5, respectively). The test was administered over 10 minutes with visual stimuli appearing randomly at variable intervals of 2 to 10 seconds. Subjects were instructed to respond to the appearance of a visual stimulus on a computer screen by pushing a response button as quickly as possible. Lapses were measured as (RT > 500 msec).
Time Frame: 2 hours post-dose
Measure: Least Squares Mean (Standard Error); unit: lapses
Arm/Group | Placebo | JZP-110
Number analyzed (Participants) | 22 | 22
lapses | 7.47 (2.357) | 3.04 (2.357)
Statistical Analysis 1: Comparison: Placebo vs JZP-110; Test type: Superiority; p = 0.0939, ANOVA

20. Secondary Outcome: PVT Number of Lapses at 6 Hours Post-dose
Description: as for outcome 19
Time Frame: 6 hours post-dose
Measure: Least Squares Mean (Standard Error); unit: lapses
Arm/Group | Placebo | JZP-110
Number analyzed (Participants) | 22 | 22
lapses | 9.88 (2.357) | 3.81 (2.357)
Statistical Analysis 1: Comparison: Placebo vs JZP-110; Test type: Superiority; p = 0.0246, ANOVA

21. Secondary Outcome: PVT Mean Reaction Time at 2 Hours Post-dose
Description: The PVT was administered at screening for practice only, and at predose and within 30 minutes before each driving test on Days 7 and 14 (Visits 4 and 5, respectively). The test was administered over 10 minutes with visual stimuli appearing randomly at variable intervals of 2 to 10 seconds. Subjects were instructed to respond to the appearance of a visual stimulus on a computer screen by pushing a response button as quickly as possible. Mean RT is measured in msec.
Time Frame: 2 hours post-dose
Measure: Least Squares Mean (Standard Error); unit: msec
Arm/Group | Placebo | JZP-110
Number analyzed (Participants) | 22 | 22
msec | 633.30 (162.286) | 311.74 (162.286)
Statistical Analysis 1: Comparison: Placebo vs JZP-110; Test type: Superiority; p = 0.1475, ANOVA

22. Secondary Outcome: PVT Mean Reaction Time at 6 Hours Post-dose
Description: as for outcome 21
Time Frame: 6 hours post-dose
Measure: Least Squares Mean (Standard Error); unit: msec
Arm/Group | Placebo | JZP-110
Number analyzed (Participants) | 22 | 22
msec | 628.26 (162.286) | 309.81 (162.286)
Statistical Analysis 1: Comparison: Placebo vs JZP-110; Test type: Superiority; p = 0.1513, ANOVA

23. Secondary Outcome: PVT Inverse Reaction Time at 2 Hours Post-dose
Description: The PVT was administered at screening for practice only, and at predose and within 30 minutes before each driving test on Days 7 and 14 (Visits 4 and 5, respectively). The test was administered over 10 minutes with visual stimuli appearing randomly at variable intervals of 2 to 10 seconds. Subjects were instructed to respond to the appearance of a visual stimulus on a computer screen by pushing a response button as quickly as possible. Inverse reaction time was expressed as 1/reaction time in msec.
Time Frame: 2 hours post-dose
Measure: Least Squares Mean (Standard Error); unit: 1/RT(ms))
Arm/Group | Placebo | JZP-110
Number analyzed (Participants) | 22 | 22
1/RT(ms)) | 3.36 (0.136) | 3.82 (0.136)
Statistical Analysis 1: Comparison: Placebo vs JZP-110; Test type: Superiority; p = 0.0002, ANOVA

24. Secondary Outcome: PVT Inverse Reaction Time at 6 Hours Post-dose
Description: as for outcome 23
Time Frame: 6 hours post-dose
Measure: Least Squares Mean (Standard Error); unit: 1/RT(ms))
Arm/Group | Placebo | JZP-110
Number analyzed (Participants) | 22 | 22
1/RT(ms)) | 3.34 (0.136) | 3.77 (0.136)
Statistical Analysis 1: Comparison: Placebo vs JZP-110; Test type: Superiority; p = 0.0005, ANOVA

25. Secondary Outcome: PVT Number of Errors of Commission at 2 Hours Post-dose
Description: The PVT was administered at screening for practice only, and at predose and within 30 minutes before each driving test on Days 7 and 14 (Visits 4 and 5, respectively). The test was administered over 10 minutes with visual stimuli appearing randomly at variable intervals of 2 to 10 seconds. Subjects were instructed to respond to the appearance of a visual stimulus on a computer screen by pushing a response button as quickly as possible. Errors of commission were measured as the number of responses without a stimulus or false starts with (RT < 100 msec).
Time Frame: 2 hours post-dose
Measure: Least Squares Mean (Standard Error); unit: errors
Arm/Group | Placebo | JZP-110
Number analyzed (Participants) | 22 | 22
errors | 1.65 (0.439) | 1.26 (0.439)
Statistical Analysis 1: Comparison: Placebo vs JZP-110; Test type: Superiority; p = 0.4774, ANOVA

26. Secondary Outcome: PVT Number of Errors of Commission at 6 Hours Post-dose
Description: as for outcome 25
Time Frame: 6 hours post-dose
Measure: Least Squares Mean (Standard Error); unit: errors
Arm/Group | Placebo | JZP-110
Number analyzed (Participants) | 22 | 22
errors | 1.92 (0.439) | 1.45 (0.439)
Statistical Analysis 1: Comparison: Placebo vs JZP-110; Test type: Superiority; p = 0.3801, ANOVA

27. Secondary Outcome: Toronto Hospital Alert Test (THAT)
Description: THAT is a 10-item self-report questionnaire designed to measure perceived alertness in the preceding week. The THAT was administered at baseline and the end of each treatment period. The total score of THAT can range between 0 to 50 where the higher score indicates greater alertness.
Time Frame: Post Treatment at day 21
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | JZP-110
Number analyzed (Participants) | 22 | 22
score on a scale | 26.83 (1.400) | 33.97 (1.397)
Statistical Analysis 1: Comparison: Placebo vs JZP-110; Test type: Superiority; p < 0.0001, ANOVA

ADVERSE EVENTS:
Time Frame: Adverse events were reported from the time written informed consent was obtained until the final study visit or early termination, up to 21 days.
Description: The Safety Population consisted of all subjects who received at least 1 dose of study medication. A treatment-emergent AE (TEAE), was defined as an AE that either began after first study drug dose or worsened after the first dose. When determining the percent of subjects who experienced an AE, multiple increases in severity were counted as one AE.
Groups:
- Placebo: Subjects received a single oral daily dose of placebo for 7 days.
- JZP-110: Subjects received a single oral daily dose of JZP-110 (150 mg/day for 3 days) then JZP-110 (300 mg/day for 4 days)
Arm/Group | Placebo | JZP-110
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 6/23 | 17/23
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=23) | JZP-110 (N=23)
Palpitations (Cardiac disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 3 (3) | 4 (4)
Somnolence (Nervous system disorders) | 2 (2) | 3 (3)
Sleep disorder (Nervous system disorders) | 1 (1) | 3 (3)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Agitation (Psychiatric disorders) | 0 (0) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review trial results communications prior to public release and can embargo such communications for a period of at least 60 days from the time submitted to sponsor for review. If requested by sponsor, the PI will withhold publication for up to an additional 30 days. Furthermore, the first publication of study results must be a joint publication of all study sites unless a joint manuscript has not been submitted for publication within 12 months of completion of the study.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-08-09): https://cdn.clinicaltrials.gov/large-docs/08/NCT02806908/SAP_000.pdf
  • Study Protocol (2018-02-07): https://cdn.clinicaltrials.gov/large-docs/08/NCT02806908/Prot_001.pdf